CLINICAL TRIAL: NCT00509613
Title: Phase 1 Dose Escalation Study With Sorafenib in Combination With Sirolimus in Patients With Solid Tumor
Brief Title: Phase 1 Study With Sorafenib and Sirolimus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: C.M.L. van Herpen, University Medical Centre Nijmegen, st Radboud
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UMCNONCO 2006_01; 2006-006454-10
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Advanced Solid Tumor; Refractory to Standard Therapies
MeSH Terms: interventions — Sorafenib; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sorafenib
Drug: Sirolimus

SUMMARY:
The purpose of the trial is to identify the recommended dose of sorafenib and sirolimus for combination therapy in subsequent phase 2 trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological or cytological confirmed advanced solid tumor, which is refractory to standard therapies or for which no standard therapy exists and for which there is a rationale for the therapeutic use of a combination of sorafenib and sirolimus (especially metastic RCC, malignant melanoma, HCC, NSCLC, pancreatic cancer, hormone refractory prostate cancer).
* Men or women of at least 18 years
* Patients who have an ECOG status of 0 or 1
* Patients who have a life expectancy of at least 12 weeks
* Adequate bone marrow, liver and renal function
* Negative pregnancy test for female patients of childbearing potential
* Women and men enrolled into this trial must use adequate birth control measures during the course of the trial.
* Signed informed consent

Exclusion Criteria:

* History of serious cardiac disease
* Active clinically serious bacterial, viral or fungal infections (> grade 2).
* Known history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C.
* Clinically symptomatic brain or meningeal metastasis.
* Patients with seizure disorders requiring medication (such as steroids or antiepileptics).
* Patients with evidence or history of bleeding diathesis.
* Substance abuse, medical, psychological or social conditions that may interfere with the patients participation in the study or evaluation of the study results.
* Concomitant treatment with strong CYP3A4 inductors (such as rifampicin, St. John´s Wort) or CYP3A4 inhibitors (such as ketoconazole, voriconazole, itraconazole, diltiazem, verapamil, erythromycin). Moderate or weak CYP3A4 modifiers should be used concomitantly only after careful assessment of risk-benefit ratio. Concomitant use of carbamazepine, phenobarbital, phenytoin or chronic use of dexamethasone is excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-06; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
identify the recommended doses for the combination of sorafenib and sirolimus for subsequent phase II studies

SECONDARY OUTCOMES:
to determine the safety profile of the combination therapy of sorafenib with sirolimus
to determine, if possible, the Maximum Tolerated Dose (MTD) of sorafenib and sirolimus in combination therapy
to analyze pharmacokinetic PK profiles (AUC, Cmax) during combination therapy for sorafenib and sirolimus
to evaluate efficacy of the combination descriptively (response rate and rate of stable diseases)

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, MD, PhD, Principal Investigator — UMC St Radboud
Locations (1):
- UMC St Radboud, Nijmegen, Netherlands